CLINICAL TRIAL: NCT04179461
Title: Personalized Treatment Algorithms for Difficult-to-treat Asthma: Bench to Community
Brief Title: Personalized Treatment Algorithms for Difficult-to-treat Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Theresa Guilbert, MD, Principal Investigator, Children's Hospital Medical Center, Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARC 7
Record Dates: First submitted 2019-11-14; First posted 2019-11-27 (Actual); Results first posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-07

CONDITIONS: Asthma in Children
MeSH Terms: interventions — Cholecalciferol; Vitamin D; Histamine Antagonists; Cetirizine; Loratadine; Azithromycin; Fluticasone; Mometasone Furoate; Formoterol Fumarate; Fluticasone-Salmeterol Drug Combination; Beclomethasone; Budesonide, Formoterol Fumarate Drug Combination; Tiotropium Bromide

STUDY DESIGN:
Intervention Model Description: The study has 3 study phases: baseline, intervention, and observation. Each participant will independently transition through these study phases.
  Baseline period: Each participant will be given a treatment recommendation according to their asthma severity/control using the National Asthma Education and Prevention Program (NAEPP asthma guidelines).
  Intervention period: Each participant will be given a personalized treatment plan based on their asthma severity/control during the baseline period, biologic, and environmental factors.
  Observation period: All participants will be observed for at least 6 months. Investigators will track the participant's personal outcomes (comparing to baseline) for reutilization, symptom-free days, and quality of life.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Personalized Treatment (Experimental): Personalized asthma treatment plan based off of individual's asthma severity/control, personal and family medical history, history of environmental exposures, adherence, medical visits, biomarker assays, and home trigger assessment.
  Study participants were prescribed recommended medications for the treatment of their asthma. These medications were prescribed through their insurance based of the of personalized treatment plan recommendation. Asthma controller medications may be increased based off of the participant's asthma control and the recommendation of the personalized plan. They would receive one of the asthma controller medications listed in the intervention.
  Interventions: Drug: Cholecalciferol; Drug: antihistamine; Drug: Azithromycin; Drug: emollient cream; Drug: Fluticasone Propionate; Drug: Asthma Controller Medication

INTERVENTIONS:
Drug: Cholecalciferol — Oral administration
  Other Names: Vitamin D
Drug: antihistamine — Oral administration
  Other Names: cetirizine; loratadine
Drug: Azithromycin — Oral administration
  Other Names: Zithromax
Drug: emollient cream — Topical
Drug: Fluticasone Propionate — Nasal spray
  Other Names: Flonase Nasal Spray
Drug: Asthma Controller Medication — Study participants asthma controller medication may be increased based off of their asthma control and the recommendation of the personalized plan.
  Other Names: Mometasone/Formoterol; Fluticasone/Salmeterol; Mometasone Furoate; Fluticasone; Beclomethasone; Budesonide/Formoterol; Tiotropium

SUMMARY:
Asthma is a common, complex and costly chronic condition. Moreover, asthma is heterogeneous in terms of treatment response. This heterogeneity contributes to the difficulty in both studying and treating asthma. This is a pilot study to improve health outcomes in youths with difficult to treat asthma with ongoing symptoms and healthcare utilization despite medium to high doses of inhaled corticosteroids. Asthma heterogeneity in both disease pathophysiology and treatment response contributes to the difficulty in both studying and managing asthma. In order to begin to develop personalized algorithms for patients, investigators need to model novel biomarkers and other factors that contribute to individual differences in asthma outcome and test other factors that contribute to individual differences in asthma outcome and test personalized treatment strategies.

DETAILED DESCRIPTION:
With this study investigators will conduct study visits to determine and quantify known molecular, genetic, genomic, epigenetics, immunologic, and exposure biomarkers that will help elucidate molecular disease endotype within the difficult-to-treat phenotype. This information will be used along with clinical, psychosocial, and adherence data to develop a personalized treatment plan. Following the personalized treatment plan, study clinicians will prescribe the medications through a home delivery or routine pharmacy depending on the family's preference and covered by the participant's health insurance. Investigators will track disease outcome metrics including exacerbations, symptom-free days, and asthma symptom scores to determine the effectiveness of this personalized approach.

ELIGIBILITY:
Inclusion Criteria:

* History of provider-diagnosed asthma
* Meets one of the following definition for NAEPP guidelines uncontrolled moderate persistent asthma or severe persistent asthma in the past 12 months:

  * NAEPP step 3-4 with one of the following criteria in the past 12 months:

    * Two Asthma Control Test (ACT) scores <20
    * 1 Urgent Care or Emergency Department visit or hospitalization for asthma
    * >2 prednisone bursts
  * NAEPP step 5-6
* Current health insurance coverage at enrollment. This will be verified at V1 at the registration desk. If the family loses insurance during the study, the patient will be referred to the pulmonary social worker and financial office for assistance
* Reside at a primary home on average 5 out of 7 days a week.
* Primary home is within a 40 mile radius of Cincinnati Children's Base location or PI's discretion.

Exclusion Criteria:

* Received biologic therapy 6 months prior to enrollment
* Received systemic steroids 6 weeks prior to enrollment
* Active chronic disease apart from asthma or allergic disease
* Co-morbid lung disease
* Dependence on immunosuppressive drugs for a condition other than asthma
* Participant is pregnant
* Has a severe bleeding disorder
* Has significant developmental disability
* Share a bedroom with a currently enrolled Breath Warriors study participant

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Guilbert, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Gurjit K Khurana Hershey, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guilbert TW, Biagini JM, Ramsey RR, Keidel K, Curtsinger K, Kroner JW, Durrani SR, Stevens M, Pilipenko V, Martin LJ, Kercsmar CM, Hommel K, Hershey GKK. Treatment by biomarker-informed endotype vs guideline care in children with difficult-to-treat asthma. Ann Allergy Asthma Immunol. 2022 May;128(5):535-543.e6. doi: 10.1016/j.anai.2022.01.030. Epub 2022 Feb 3. PMID 35123074

RESULTS

PARTICIPANT FLOW:
Groups:
- Personalized Treatment: Personalized asthma treatment plan based off of individual's asthma severity/control, personal and family medical history, history of environmental exposures, adherence, medical visits, biomarker assays, and home trigger assessment.
  Study participants were prescribed recommended medications for the treatment of their asthma. These medications were prescribed through their insurance based of the of personalized treatment plan recommendation. Asthma controller medications may be increased based off of the participant's asthma control and the recommendation of the personalized plan. They would receive one of the asthma controller medications listed in the intervention.
  Cholecalciferol: Oral administration
  antihistamine: Oral administration
  Azithromycin: Oral administration
  emollient cream: Topical
  Fluticasone Propionate: Nasal spray
  Asthma Controller Medication: Study participants asthma controller medication may be increased based off of their asthma control and the recommendation of the personalized plan.
Period: Overall Study
Arm/Group | Personalized Treatment
Started | 21
Completed | 17
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: 1 participant withdrew from the study prior to being assigned a personalized treatment.
Arm/Group | Personalized Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Primary home within a 40 mile radius of Cincinnati Children's Base Location [Count of Participants; unit: Participants] | 20
Health insurance coverage at enrollment [Count of Participants; unit: Participants] | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Composite Asthma Severity Index (CASI)
Description: CASI was measured by questionnaire and is a severity score of symptom burden, exacerbations, healthcare utilization, lung function and dose of inhaled corticosteroids. The change in CASI score was calculated between V1 (Baseline), V2 (Guideline Care - before intervention), and V3 (12 Months).
  [The CASI score has a minimum value = 0, maximum value = 20, a higher score indicates greater asthma severity]
Time Frame: Baseline to 12 months
Population: 17 participants whom had complete data sets were analyzed. 4 participants withdrew early from the study and were not included in this analysis due to incomplete data.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Personalized Treatment
Number analyzed (Participants) | 17
score on a scale
  V1 | 5 [5 to 6]
  V2 | 5 [5 to 5]
  V3 | 5 [5 to 5]
Statistical Analysis 1: Comparison: Personalized Treatment; The modified CASI score incorporates key asthma outcomes such as symptoms, healthcare utilization, and medication dose; Test type: Equivalence — The Wilcoxon signed-rank test was employed for pairwise comparison between visits for continuous data. Data for the CASI was captured at clinical visits. 3. A level of statistical significance was established at < 0.05; p = 0.52, Wilcoxon (Mann-Whitney) — Change in CASI score from V1 to V3

2. Secondary Outcome: Asthma Control Test (ACT)
Description: ACT was measured by questionnaire, assessing frequency of reported asthma symptoms, rescue medication use, the effect of asthma on daily functioning, and overall asthma control. The change in ACT score was calculated between V1 (Baseline), V2 (Guideline Care - before intervention), and V3 (12 Months).
  [The ACT score has a minimum value = 5, maximum value = 25, a score 19 indicates well-controlled asthma]
Time Frame: Baseline to 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Personalized Treatment
Number analyzed (Participants) | 17
score on a scale
  V1 | 23.0 [20.0 to 23.0]
  V2 | 21.7 [18.2 to 24.2]
  V3 | 22.5 [18.2 to 24.2]
Statistical Analysis 1: Comparison: Personalized Treatment; Test type: Equivalence — The Wilcoxon signed-rank test was employed for pairwise comparison between visits for continuous data. Data for the c-ACT/ACT was captured at clinical visits and from monthly phone calls. Because c-ACT/ACT could vary through time, we calculated the average c-ACT/ACT between V1-V2 and V2-V3. Data analysis was performed in SAS version 9.4 (SAS, Cary, NC). A level of statistical significance was established at < 0.05; p = 0.45, Wilcoxon (Mann-Whitney) — The change in ACT score from V1 to V2 (the period between V1 and V2)
Statistical Analysis 2: Comparison: Personalized Treatment; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.01, Wilcoxon (Mann-Whitney) — The change in ACT score from V1-V2 to V2-V3

3. Secondary Outcome: Pulmonary Function Measured by Spirometry: Forced Expiratory Volume in 1 Second (FEV1) / Forced Vital Capacity (FVC)
Description: FEV1 is air volume exhaled in 1 second during spirometry. Forced vital capacity is the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. The change in FEV1/FVC was calculated between V1 (Baseline), V2 (Guideline Care - before intervention), and V3 (12 Months). This will be used as a measurement in asthma severity.
  [A lower FEV1/FVC ratio indicates more severe asthma]
Time Frame: Baseline to 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Personalized Treatment
Number analyzed (Participants) | 17
Ratio
  V1 | 0.81 [0.76 to 0.86]
  V2 | 0.8 [0.76 to 0.85]
  V3 | 0.8 [0.77 to 0.87]
Statistical Analysis 1: Comparison: Personalized Treatment; Test type: Equivalence — The Wilcoxon signed-rank test was employed for pairwise comparison between visits for continuous data and the Bowker's test was used to compare categorical FEV1-FVC data. Data analysis was performed in SAS version 9.4 (SAS, Cary, NC). A level of statistical significance was established at < 0.05; p = 0.27, Wilcoxon (Mann-Whitney) — The Change in FEV1/FVC from Visit 1 to Visit 3

4. Secondary Outcome: Adherence of Asthma Controller Medication
Description: Adherence was measured using the Propeller Health Inhaler monitor and web-based software management platform that tracks adherence of asthma medications. The change in adherence was calculated between V1 (baseline) to V3 (12 Months).
Time Frame: Baseline to 12 months
Population: 16 participants whom had complete data sets were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentage of medication taken
Arm/Group | Personalized Treatment
Number analyzed (Participants) | 16
percentage of medication taken
  V1 | 42 [21 to 57]
  V3 | 36 [14 to 53]
Statistical Analysis 1: Comparison: Personalized Treatment; Test type: Equivalence — Intervention adherence and end of study adherence were each calculated based on the 30 days prior to end of intervention and V3, respectively, in order to assess a consistent timeframe. The paired Wilcoxon signed rank test was conducted to compare controller inhaler adherence during baseline, adherence intervention, and end of study; p = 0.17, Wilcoxon (Mann-Whitney) — Change between baseline (V1) to end of study (V3)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Review for possible adverse events was completed at study visits and follow-up phone calls by the research coordinator. If adverse events were identified, they were documented on the Adverse Event Reporting Form and reviewed at the meeting of the Steering committee.
Arm/Group | Personalized Treatment
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 12/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Personalized Treatment (N=21)
Major Depressive Disorder (Psychiatric disorders) | 1 (1) — Major depressive disorder requiring hospitalization
Psychiatric Evaluation (Psychiatric disorders) | 1 (2) — Psychiatric Evaluation requiring hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Personalized Treatment (N=21)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 8 (12)
Ankle Injury (Musculoskeletal and connective tissue disorders) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Streptococcal Pharyngitis (Infections and infestations) | 3 (3)
Viral Gastroenteritis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT04179461/Prot_SAP_000.pdf